CLINICAL TRIAL: NCT07353723
Title: A Pilot Study to Assess Feasibility and Preliminary Efficacy of Neoadjuvant Nimotuzumab, Toripalimab, and Chemotherapy in Locally Advanced Tonsillar Cancer
Brief Title: Nimotuzumab Combined With Toripalimab and Chemotherapy for Locally Advanced Tonsillar Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025HNST01
Record Dates: First submitted 2025-12-22; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Head & Neck Cancer
Keywords: Nimotuzumab; neouAdjuvant; pathological complete response, pCR
MeSH Terms: conditions — Head and Neck Neoplasms; Pathologic Complete Response | interventions — nimotuzumab; toripalimab; 130-nm albumin-bound paclitaxel; Carboplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab Combined with Toripalimab and Chemotherapy (Experimental): treatment Regimens:Nimotuzumab 400 mg, intravenous infusion(IV), d1, Q3W, for 2 cycles;Nab-paclitaxel 260 mg/m², intravenous infusion(IV), d1, Q3W,for 2 -4cycles; Carboplatin dosage was calculated using the Calvert formula (dose = target AUC × [GFR + 25]), d1,IV,Q3W,for 2-4 cycles. Toripalimab 240 mg, IV,d1, Q3W, for 2-4 cycles.Each infusion should be given over at least 60 minutes, with close monitoring for infusion-related reactions.All patients received 2 -4cycles of neoadjuvant combination therapy, followed by endoscopy combined with imaging evaluation around Day 42.
  Interventions: Drug: Nimotuzumab; Drug: Toripalimab; Drug: Nab-paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: Nimotuzumab — treatment Regimen:Nimotuzumab was administered by intravenous infusion at a dose of 400 mg,d1, Q3W,for 2-4 cycles
  Other Name:
  Other Names: Nimotuzumab Injection
Drug: Toripalimab — treatment Regimen:Toripalimab was administered by intravenous infusion at a dose of 240 mg,d1,Q3W,for 2-4 cycles
Drug: Nab-paclitaxel — treatment Regimen:Nab-paclitaxel was administered by intravenous infusion at a dose of 260mg/m² ,d1, Q3W,for 2-4 cycles
Drug: carboplatin — treatment Regimen: Carboplatin dosage was calculated using the Calvert formula (dose = target AUC × [GFR + 25]), d1,IV,Q3W,for 2-4 cycles
  Other Names: Carboplatin (neoadjuvant）; Carboplatin (AUC 6); Carboplatin (AUC 5)

SUMMARY:
This is a prospective,single-arm,Phase II clinical study to designed to evaluate the efficancy and safety of nimotuzumab Combined with Toripalimab and Chemotherapy for Locally Advanced Tonsillar Cancer

DETAILED DESCRIPTION:
This study is a prospective,single-arm,Phase II clinical study to evaluate the efficancy and safety of nimotuzumab Combined with Toripalimab and Chemotherapy for Locally Advanced Tonsillar Cancer,The study aims to explore whether nimotuzumab Combined with Toripalimab and Chemotherapy for Locally Advanced Tonsillar Cancer, can improve the pathological complete response (pCR) and overall survival rate(OS) compared with the historical data. The study plans to enroll approximately 10 patients at Tangdu Hospital and expected to completed enrollment within 1 yeasrs,within an additional 5 years follow-up for the label-enrolled subject.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old (inclusive of 18 and 80 years), of either gender.
2. Histopathologically or cytologically confirmed, and diagnosed as resectable locally advanced tonsillar squamous cell carcinoma (TSCC) by MRI imaging.
3. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
4. Male subjects are eligible if they agree to comply with the following standards during treatment and for at least 180 days after the last cycle of chemotherapy:a) Prohibition of sperm donation;AND• Abstain from heterosexual intercourse as a usual and preferred lifestyle (long-term and persistent abstinence) and agree to maintain abstinence;OR• Agree to use contraceptive measures unless confirmed as azoospermic (vasectomy or secondary to medical reasons, see Appendix 5), with details as follows:→ Use a male condom during penile-vaginal intercourse with a reproductive-aged female partner who is not currently pregnant, and the partner uses an additional contraceptive method.Note: Males whose partners are pregnant or breastfeeding must agree to either maintain abstinence from penile-vaginal intercourse at all times or use a male condom for every penile-vaginal penetration.b) Male subjects must also agree to use a male condom during any activity that allows ejaculation with others of any gender.c) Contraceptive methods used by males must comply with regulations regarding contraception in clinical research participation.
5. Female subjects are eligible if they are not pregnant or breastfeeding, and meet at least one of the following conditions:(1) Not a woman of childbearing potential (WOCBP);OR(2) If a WOCBP, use a highly effective contraceptive method (annual failure rate <1%) with low user dependence, or abstain from heterosexual intercourse as a preferred and regular lifestyle (long-term and persistent abstinence) during the intervention period and for at least 210 days after the last cycle of chemotherapy, and agree not to donate ova (eggs, oocytes) to others or freeze/store ova for personal reproductive purposes during this period. Investigators shall evaluate the likelihood of contraceptive method failure (i.e., non-compliance, recent initiation) relative to the first administration of study treatment.a) WOCBP must have a negative result on a highly sensitive urine or serum pregnancy test (urine or serum test selected per regulatory requirements) within 24 hours (urine) or 72 hours (serum) before the first administration of study treatment to be enrolled.Note: If the interval between the screening pregnancy test and the first administration of study intervention exceeds 24 hours (urine) or 72 hours (serum), a repeat pregnancy test (urine or serum) must be performed, and the result must be negative for the subject to start receiving study medication.b) If a urine test is inconclusive (e.g., unclear result), a serum pregnancy test is required. In such cases, subjects with a positive serum pregnancy test result must be excluded.c) Investigators are responsible for reviewing medical history, menstrual history, and recent sexual activity to reduce the risk of enrolling women with undetected early pregnancy.d) Contraceptive methods used by females must comply with regulations regarding contraception in clinical research participation;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2 within 3 days before the first administration of study intervention.
7. Evidence of extranodal extension (ENE) in lymph nodes (confirmed by MRI, CT, or pathology).
8. Voluntarily sign the written informed consent form for the study.
9. Expected survival time ≥6 months.
10. Adequate organ function as indicated by screening laboratory test results.a) Hematological parameters:White blood cell (WBC) count ≥4 × 10⁹/L;Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L;Platelet count ≥100 × 10⁹/L;Hemoglobin (Hb) ≥90 g/L;b) Renal function:Serum creatinine ≤1.5 × upper limit of normal (ULN), or creatinine clearance (CrCl) >60 mL/min (calculated using the Cockcroft-Gault formula):Female: CrCl = [(140 - age) × body weight (kg) × 0.85] / (72 × Scr [mg/dL])Male: CrCl = [(140 - age) × body weight (kg) × 1.00] / (72 × Scr [mg/dL])c) Hepatic function:Serum total bilirubin ≤1.5 × ULN;Aspartate aminotransferase (AST) ≤2.5 × ULN;Alanine aminotransferase (ALT) ≤2.5 × ULN;d) Coagulation function:International Normalized Ratio (INR) ≤1.5;Prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤1.5 × ULN.
11. Good compliance and willingness to cooperate with follow-up procedures.

Exclusion Criteria:

1. Prior systemic therapy for advanced (metastatic) or unresectable (locally advanced) tonsillar cancer, except for permitted neoadjuvant/adjuvant therapy. Neoadjuvant/adjuvant therapy must have been completed at least 6 months before the diagnosis of advanced and/or unresectable disease. Subjects who received prior neoadjuvant/adjuvant therapy and had R2 pathology after tumor resection are excluded.
2. Active autoimmune disease requiring systemic therapy (i.e., disease-modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. Replacement therapies (e.g., thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) are not considered systemic therapy and are permitted.
3. Major surgery prior to the initiation of study intervention with inadequate recovery from surgery and/or surgical complications.
4. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or drugs targeting other stimulatory or co-inhibitory T-cell receptors (e.g., CTLA-4, OX-40, CD137).
5. Prior treatment with EGFR-targeted agents.
6. Anti-tumor therapy for advanced tonsillar cancer, including investigational drugs, within 4 weeks before enrollment.
7. Unresolved adverse events (AEs) from prior anti-cancer therapy (i.e., AEs > Grade 1 or baseline). Subjects with neuropathy ≤ Grade 2 may be eligible based on investigator assessment.
8. Radiotherapy within 2 weeks before the start of investigational treatment. Subjects must have recovered from all radiotherapy-related toxicities, be free of corticosteroid use, and have no history of radiation pneumonitis. A 1-week washout period is permitted for palliative radiotherapy (≤2 weeks of radiotherapy) for non-central nervous system (CNS) disease (if deemed safe by the investigator). A 2-week washout period is required for longer radiotherapy courses (>2 weeks).
9. Administration of live vaccines within 30 days before the first dose of study drug.Note: Live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, bacillus Calmette-Guérin (BCG), and typhoid vaccines. Seasonal influenza vaccines administered by injection are generally inactivated virus vaccines and are permitted; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not permitted.
10. Current or prior participation in a study of an investigational drug, or use of an investigational device within 4 weeks before the first dose of study drug.Note: Subjects who have entered the follow-up phase of an investigational study are eligible to participate in this study if at least 4 weeks have passed since the last dose of the prior investigational drug.
11. Diagnosis of immunodeficiency or receipt of long-term systemic corticosteroid therapy (dose exceeding 10 mg prednisone equivalent per day) or any form of immunosuppressive therapy within 7 days before the first dose of study drug.
12. History of another invasive malignancy that is progressive or required active treatment within the past 3 years.Note: Subjects with a history of skin basal cell carcinoma, skin squamous cell carcinoma, or carcinoma in situ (e.g., ductal carcinoma in situ of the breast, cervical carcinoma in situ) who have received potentially curative treatment are not excluded.
13. Severe hypersensitivity reaction (> Grade 3) to toripalimab, nimotuzumab, albumin-bound paclitaxel, carboplatin, and/or any of their excipients.
14. History of (non-infectious) pneumonitis requiring corticosteroid therapy, or current pneumonitis.
15. Active infection requiring systemic therapy.
16. Known history of human immunodeficiency virus (HIV) infection.
17. Known active tuberculosis (TB; Mycobacterium tuberculosis).
18. Severe, poorly controlled concurrent diseases (e.g., heart failure, diabetes mellitus, hypertension, liver failure, renal failure, thyroid disease, psychiatric illness, etc.).
19. Major surgery within 30 days before the first dose of investigational drug or planned surgery during the study period.
20. Inappropriate for study participation as assessed by the investigator.
21. Unwillingness to participate in the study or inability to sign the informed consent form.
22. Known history or any evidence of central nervous system (CNS) metastases and/or carcinomatous meningitis as assessed by the study site investigator.
23. History or evidence of disease, treatment, or abnormal laboratory values that may interfere with trial results, prevent full participation in the study (e.g., hearing impairment), or that the investigator believes would not be in the subject's best interest to participate.
24. Known psychiatric illness or substance abuse disorder that would interfere with the subject's ability to comply with study requirements.
25. History of allogeneic tissue/solid organ transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | Within 1-2 week after radical surgery (same time point as MPR assessment)
  no residual tumor cells in the primary lesion and lymph nodes after surgery (pathological assessment).

SECONDARY OUTCOMES:
Surgical resection margin (first margin and second margin) | Within 1-2 week after radical surgery (performed 2-3 weeks after the completion of 2 cycles of neoadjuvant treatment)
  First margin: tumor margin before neoadjuvant therapy;
  Second margin: tumor margin after neoadjuvant therapy (defined as Clear margin per the 2025 NCCN Guidelines: the distance from invasive tumor to the resection margin ≥ 5 mm).
Major pathological response rate (MPR) | Within 1-2 week after radical surgery (performed 2-3 weeks after the completion of 2 cycles of neoadjuvant treatment)
  residual tumor in the primary lesion < 10% (pathological assessment).
Radiological response rate | After the completion of 2 cycles of neoadjuvant treatment (each cycle is 21 days)
  evaluated by contrast-enhanced CT/MRI before and after treatment (per RECIST 1.1 criteria: complete response [CR]/partial response [PR]/stable disease [SD]/progressive disease [PD]).
Functional preservation rate | functional assessment: before surgery,and 1 month, 6 months, and 1 year after surgery or Concurrent chemoradiotherapy
  Functional preservation rate was defined as the proportion of patients with normal phonation and swallowing function: before surgery, and 1 month, 6 months, and 1 year after surgery or radiotherapy (evaluated via video laryngoscopy + scale assessment + voice analysis)
Disease-free survival (DFS) | 72 months after treatment initiation
  the time from the initiation of radical treatment to the first occurrence of disease recurrence, metastasis, second primary cancer, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao DaQing, Principal Investigator — Tangdu Hospital, Air Force Medical University (AFMU), Xi'an, China
Locations (1):
- Tangdu Hospital, Air Force Medical University, Xi'an 710038, Shaanxi Province, China, Shanxi, Province, China

IPD SHARING:
Plan to Share IPD: No